CLINICAL TRIAL: NCT03067441
Title: A Multicenter Open-Label Extension (OLE) Study To Assess The Long-Term Safety and Efficacy of Bempedoic Acid (ETC-1002) 180 MG
Brief Title: Assessment of the Long-Term Safety and Efficacy of Bempedoic Acid (CLEAR Harmony OLE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1002-050; 2016-004115-12 (EudraCT Number)
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia; Atherosclerotic Cardiovascular Disease
Keywords: hyperlipidemia; cholesterol; heterozygous familial hypercholesterolemia; atherosclerotic cardiovascular disease; ASCVD; HeFH; LDL
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis; Hyperlipidemias | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label bempedoic acid (Experimental): bempedoic acid 180 mg tablet
  Interventions: Drug: bempedoic acid

INTERVENTIONS:
Drug: bempedoic acid — bempedoic acid 180 mg tablets taken orally, once per day.
  Other Names: ETC-1002

SUMMARY:
The purpose of this study is to see if bempedoic acid (ETC-1002) is safe and well-tolerated in patients with high cardiovascular risk and elevated LDL cholesterol that is not adequately controlled by their current therapy.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed CLEAR Harmony (1002-040) parent study

Exclusion Criteria:

* Experienced a treatment-related SAE that led to study drug discontinuation in the CLEAR Harmony (1002-040) parent study.
* Medical condition requires lipid measurement and/or adjustment of background lipid-regulating therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1462 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Esperion Therapeutics, Inc.
Locations (3):
- United States (3):
  - Jedidiah Clinical Research, Tampa, Florida
  - L-MARC Research Center, Louisville, Kentucky
  - Sentral Clinical Research Services, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] Goldberg AC, Hopkins PN, Toth PP, Ballantyne CM, Rader DJ, Robinson JG, Daniels SR, Gidding SS, de Ferranti SD, Ito MK, McGowan MP, Moriarty PM, Cromwell WC, Ross JL, Ziajka PE; National Lipid Association Expert Panel on Familial Hypercholesterolemia. Familial hypercholesterolemia: screening, diagnosis and management of pediatric and adult patients: clinical guidance from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Clin Lipidol. 2011 Jun;5(3 Suppl):S1-8. doi: 10.1016/j.jacl.2011.04.003. Epub 2011 Apr 12. PMID 21600525
- [Background] Pollex RL, Joy TR, Hegele RA. Emerging antidyslipidemic drugs. Expert Opin Emerg Drugs. 2008 Jun;13(2):363-81. doi: 10.1517/14728214.13.2.363. PMID 18537526
- [Background] Sharrett AR, Ballantyne CM, Coady SA, Heiss G, Sorlie PD, Catellier D, Patsch W; Atherosclerosis Risk in Communities Study Group. Coronary heart disease prediction from lipoprotein cholesterol levels, triglycerides, lipoprotein(a), apolipoproteins A-I and B, and HDL density subfractions: The Atherosclerosis Risk in Communities (ARIC) Study. Circulation. 2001 Sep 4;104(10):1108-13. doi: 10.1161/hc3501.095214. PMID 11535564
- See also: World Health Organization Fact Sheet No. 317 — http://www.who.int/mediacentre/factsheets/fs317/en/
- See also: Familial Hypercholesterolemia Foundation — https://thefhfoundation.org/about-fh/what-is-familial-hypercholesterolemia
- See also: National Organization for Rare Disorders - Familial Hypercholesterolemia — https://rarediseases.org/rare-diseases/familial-hypercholesterolemia/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After successfully completing 52 weeks of treatment in the parent study, Study 1002-040 (NCT02666664), and meeting entry criteria, participants could enrol into this Open-label Extension (OLE) study.
Groups:
- Placebo; Bempedoic Acid: In the parent study (Study 1002-040), participants received placebo tablet, once daily by mouth for 52 weeks. In addition, participants received stable background lipid-modifying therapy(ies), including a maximally tolerated statin, throughout the study. Participants received open-label bempedoic acid 180 milligrams (mg) once daily by mouth for up to 78 weeks after rolling over from the parent study, followed by a 4-week period off of investigational medicinal product (IMP).
- Bempedoic Acid; Bempedoic Acid: In the parent study, participants received bempedoic acid 180 mg tablet, once daily by mouth for 52 weeks. In addition, participants received stable background lipid-modifying therapy(ies), including a maximally tolerated statin, throughout the study. Participants received open-label bempedoic acid 180 mg once daily by mouth for up to 78 weeks after rolling over from the parent study, followed by a 4-week period off of IMP.
Period: Overall Study
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid
Started | 492 | 970
Completed | 459 | 913
Not Completed | 33 | 57
Not completed — Withdrawal by Subject | 16 | 34
Not completed — Lost to Follow-up | 7 | 5
Not completed — Adverse Event | 7 | 14
Not completed — Study Terminated by Sponsor or Investigator | 1 | 0
Not completed — Physician Decision | 1 | 3
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all enrolled participants who received at least 1 dose of bempedoic acid in the Open-Label Extension (OLE) Study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | Total
Number analyzed (Participants) | 492 | 970 | 1462
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (8.54) | 66.5 (8.81) | 66.9 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 239 | 381
  Male | 350 | 731 | 1081
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 23 | 29
  White | 480 | 931 | 1411
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 3 | 4
Low-density lipoprotein cholesterol (LDL-C): Parent Study [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1)
  milligrams per deciliter (mg/dL) | 98.96 (24.171) | 102.94 (29.899) | 101.60 (28.156)
Non-high-density lipoprotein cholesterol (N-HDL-C): Parent Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 126.41 (28.531) | 130.09 (34.727) | 128.85 (32.809)
Total cholesterol: Parent Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 175.33 (30.026) | 178.94 (36.057) | 177.73 (34.179)
Apolipoprotein B: Parent Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last value prior to first dose of study drug. Population: Only participants with non-missing data were analysed.
  mg/dL
    number analyzed (Participants) | 487 | 969 | 1456
    (all) | 85.1 (19.25) | 88.2 (21.71) | 87.2 (20.97)
High-sensitivity C-reactive protein (hs-CRP): Parent Study [Median (Inter-Quartile Range); unit: milligrams per Liter (mg/L)] — Baseline was defined as the last value prior to the first dose of study drug. Population: Only participants with non-missing data were analysed.
  milligrams per Liter (mg/L)
    number analyzed (Participants) | 490 | 969 | 1459
    (all) | 1.515 [0.810 to 3.490] | 1.500 [0.700 to 3.220] | 1.510 [0.750 to 3.320]
Triglycerides: Parent Study [Median (Inter-Quartile Range); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 122.00 [97.50 to 169.25] | 125.00 [97.00 to 164.50] | 124.00 [97.50 to 166.50]
High-density lipoprotein cholesterol (HDL-C): Parent Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1).
  mg/dL | 48.93 (11.206) | 48.82 (11.790) | 48.86 (11.593)
LDL-C: OLE Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
  mg/dL | 99.5 (28.59) | 86.6 (30.18) | 91.0 (30.26)
N-HDL-C: OLE Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
  mg/dL | 126.1 (32.61) | 113.7 (34.57) | 117.9 (34.42)
Total cholesterol: OLE Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
  mg/dL | 175.2 (34.23) | 159.8 (36.41) | 165.0 (36.41)
Apolipoprotein B: OLE Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
  mg/dL | 87.6 (22.74) | 80.4 (21.31) | 82.8 (22.07)
hs-CRP: OLE Study [Median (Inter-Quartile Range); unit: mg/L] — Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
  mg/L | 1.560 [0.745 to 3.015] | 1.250 [0.620 to 2.480] | 1.325 [0.650 to 2.650]
Triglycerides: OLE Study [Median (Inter-Quartile Range); unit: mg/dL] — Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
  mg/dL | 120.0 [91.5 to 165.0] | 121.0 [88.0 to 172.0] | 120.0 [88.0 to 169.0]
HDL-C: OLE Study [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
  mg/dL | 49.0 (11.72) | 46.1 (13.00) | 47.1 (12.66)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are defined as adverse events that began or worsened in severity after the first dose of investigational medicinal product (IMP) until 30 days after the last dose in the Open-Label Extension (OLE) Study.
Time Frame: Up to Week 82
Population: Safety Population: all enrolled participants who received at least 1 dose of bempedoic acid in the OLE Study
Measure: Count of Participants; unit: Participants
Groups:
- OLE Bempedoic Acid: In the parent study, participants received either bempedoic acid 180 mg tablet or matching placebo, once daily by mouth for 52 weeks. In addition, participants received stable background lipid-modifying therapy(ies), including a maximally tolerated statin, throughout the study. Participants received open-label bempedoic acid 180 mg once daily by mouth for up to 78 weeks after rolling over from the parent study, followed by a 4-week period off of IMP.
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
Participants
  Participants with TEAEs | 385 | 758 | 1143
  Participants with serious TEAEs | 97 | 202 | 299
  Participants with TEAEs of mild severity | 93 | 195 | 288
  Participants with TEAEs of moderate severity | 211 | 403 | 614
  Participants with TEAEs of severe severity | 81 | 160 | 241

2. Secondary Outcome: Percent Change From Parent Study Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: LDL-C value at Week 52/Week 78 minus Parent Study Baseline value divided by Parent Study Baseline value multiplied by 100. Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1) in the Parent Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo; Bempedoic Acid: In the parent study (Study 1002-040), participants received placebo tablet, once daily by mouth for 52 weeks. In addition, participants received stable background lipid-modifying therapy(ies), including a maximally tolerated statin, throughout the study. Participants received open-label bempedoic acid 180 milligrams (mg) once daily by mouth for up to 78 weeks after rolling over from the parent study, followed by a 4-week period off of IMP.
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 909 | 1373
  Week 52 | -12.82 (23.419) | -13.80 (25.018) | -13.47 (24.485)
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -14.99 (23.660) | -14.15 (25.113) | -14.43 (24.632)

3. Secondary Outcome: Mean Change From Parent Study Baseline in LDL-C at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Mean change from Baseline was calculated as: Mean LDL-C value at Week 52/Week 78 minus Mean Parent Study Baseline value. Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1) in the Parent Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
milligrams per deciliter (mg/dL)
  Week 52: number analyzed (Participants) | 464 | 909 | 1373
  Week 52 | -14.08 (24.995) | -15.77 (28.123) | -15.19 (27.109)
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -16.11 (25.628) | -16.04 (28.929) | -16.06 (27.862)

4. Secondary Outcome: Percent Change From Parent Study Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: non-HDL-C value at Week 52/Week 78 minus Parent Study Baseline value divided by Parent Study Baseline value multiplied by 100. Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1) in the Parent Study.
Time Frame: Baseline; Week 52 and Week 72
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 463 | 909 | 1372
  Week 52 | -10.60 (20.722) | -10.55 (22.682) | -10.57 (22.033)
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -12.50 (22.081) | -10.82 (23.910) | -11.38 (23.321)

5. Secondary Outcome: Percent Change From Parent Study Baseline in Total Cholesterol at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: Total cholesterol value at Week 52/Week 78 minus Parent Study Baseline value divided by Parent Study Baseline value multiplied by 100. Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1) in the Parent Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 910 | 1374
  Week 52 | -9.01 (15.961) | -9.79 (16.893) | -9.53 (16.582)
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -10.15 (16.541) | -9.34 (18.030) | -9.61 (17.545)

6. Secondary Outcome: Percent Change From Parent Study Baseline in Apolipoprotein B (ApoB) at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: ApoB value at Week 52/Week 78 minus Parent Study Baseline value divided by Parent Study Baseline value multiplied by 100. Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1) in the Parent Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 458 | 905 | 1363
  Week 52 | -7.5 (20.52) | -8.8 (21.89) | -8.4 (21.44)
  Week 78: number analyzed (Participants) | 424 | 858 | 1282
  Week 78 | -7.6 (22.15) | -7.0 (22.33) | -7.2 (22.26)

7. Secondary Outcome: Percent Change From Parent Study Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP) at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: hs-CRP value at Week 52/Week 78 minus Parent Study Baseline value divided by Parent Study Baseline value multiplied by 100. Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1) in the Parent Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 462 | 908 | 1370
  Week 52 | -11.553 [-53.120 to 44.167] | -19.709 [-52.617 to 34.151] | -16.476 [-52.874 to 41.667]
  Week 78: number analyzed (Participants) | 431 | 865 | 1296
  Week 78 | -15.005 [-50.510 to 44.000] | -18.065 [-51.701 to 50.505] | -16.740 [-51.577 to 48.279]

8. Secondary Outcome: Percent Change From Parent Study Baseline in Triglycerides at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: Triglycerides value at Week 52/Week 78 minus Parent Study Baseline value divided by Parent Study Baseline value multiplied by 100. Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1) in the Parent Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 909 | 1373
  Week 52 | -4.31 [-24.08 to 21.75] | -3.21 [-22.76 to 23.50] | -3.49 [-23.02 to 22.40]
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -5.00 [-25.54 to 24.26] | -2.60 [-21.41 to 27.47] | -3.08 [-22.78 to 26.67]

9. Secondary Outcome: Percent Change From Parent Study Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: HDL-C value at Week 52/Week 78 minus Parent Study Baseline value divided by Parent Study Baseline value multiplied by 100. Baseline was defined as the mean of the values at screening and predose Day 1/Week 0 (Visit T1) in the Parent Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 907 | 1371
  Week 52 | -4.54 (16.747) | -7.06 (15.638) | -6.20 (16.060)
  Week 78: number analyzed (Participants) | 433 | 863 | 1296
  Week 78 | -3.42 (17.555) | -4.91 (16.731) | -4.41 (17.018)

10. Secondary Outcome: Percent Change From Open-Label Extension (OLE) Study Baseline in LDL-C at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: LDL-C value at Week 52/Week 78 minus OLE Study Baseline value divided by Parent Study Baseline value multiplied by 100. Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 909 | 1373
  Week 52 | -12.4 (23.79) | 3.6 (27.49) | -1.8 (27.35)
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -14.3 (25.79) | 3.7 (30.63) | -2.3 (30.31)

11. Secondary Outcome: Mean Change From OLE Baseline in LDL-C at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Mean change from Baseline was calculated as: Mean LDL-C value at Week 52/Week 78 minus Mean OLE Study Baseline value. Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
Time Frame: Baseline; Week 52 and Week 72
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
mg/dL
  Week 52: number analyzed (Participants) | 464 | 909 | 1373
  Week 52 | -14.7 (25.63) | 0.6 (24.92) | -4.6 (26.17)
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -17.0 (28.56) | 0.2 (26.04) | -5.5 (28.08)

12. Secondary Outcome: Percent Change From OLE Baseline in Non-HDL-C at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: non-HDL-C value at Week 52/Week 78 minus OLE Study Baseline value divided by OLE Study Baseline value multiplied by 100. Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 463 | 909 | 1372
  Week 52 | -10.0 (20.81) | 2.9 (23.98) | -1.4 (23.75)
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -11.8 (23.08) | 3.1 (28.02) | -1.9 (27.38)

13. Secondary Outcome: Percent Change From OLE Baseline in Total Cholesterol at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: Total Cholesterol value at Week 52/Week 78 minus OLE Study Baseline value divided by OLE Study Baseline value multiplied by 100. Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 910 | 1374
  Week 52 | -8.7 (15.78) | 1.3 (17.23) | -2.1 (17.40)
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -9.7 (17.39) | 2.1 (19.88) | -1.8 (19.88)

14. Secondary Outcome: Percent Change From OLE Baseline ApoB at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: ApoB value at Week 52/Week 78 minus OLE Study Baseline value divided by OLE Study Baseline value multiplied by 100. Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 463 | 906 | 1369
  Week 52 | -10.0 (19.94) | 0.2 (21.48) | -3.2 (21.51)
  Week 78: number analyzed (Participants) | 428 | 858 | 1286
  Week 78 | -10.2 (21.84) | 2.4 (23.16) | -1.8 (23.49)

15. Secondary Outcome: Percent Change From OLE Baseline in Hs-CRP at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: hs-CRP value at Week 52/Week 78 minus OLE Study Baseline value divided by OLE Study Baseline value multiplied by 100. Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 909 | 1373
  Week 52 | -11.720 [-50.315 to 38.433] | -2.174 [-39.583 to 61.765] | -4.856 [-43.750 to 52.800]
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -14.953 [-50.549 to 43.333] | 3.774 [-36.842 to 69.136] | -2.538 [-41.509 to 60.268]

16. Secondary Outcome: Percent Change From OLE Baseline in Triglycerides at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: Triglycerides value at Week 52/Week 78 minus OLE Study Baseline value divided by OLE Study Baseline value multiplied by 100. Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 909 | 1373
  Week 52 | 0.3 [-22.4 to 23.6] | 0.9 [-20.2 to 25.2] | 0.7 [-20.7 to 24.3]
  Week 78: number analyzed (Participants) | 433 | 865 | 1298
  Week 78 | -2.0 [-23.8 to 24.1] | 2.2 [-19.2 to 27.2] | 0.9 [-20.9 to 26.6]

17. Secondary Outcome: Percent Change From OLE Baseline in HDL-C at Weeks 52 and 78
Description: Blood samples were drawn after a minimum 10-hour fast at pre-specified intervals. Percent change from Baseline was calculated as: HDL-C value at Week 52/Week 78 minus OLE Study Baseline value divided by OLE Study Baseline value multiplied by 100. Baseline was defined as the last non-missing record prior to treatment start in the OLE Study.
Time Frame: Baseline; Week 52 and Week 78
Population: Safety Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
Number analyzed (Participants) | 492 | 970 | 1462
percent change
  Week 52: number analyzed (Participants) | 464 | 907 | 1371
  Week 52 | -4.3 (18.36) | -0.6 (14.88) | -1.8 (16.23)
  Week 78: number analyzed (Participants) | 433 | 863 | 1296
  Week 78 | -3.4 (17.77) | 2.7 (23.60) | 0.7 (22.01)

ADVERSE EVENTS:
Time Frame: Up to Week 82
Description: Treatment-emergent adverse events, defined as adverse events that began or worsened in severity after the first dose of investigational medicinal product (IMP) until 30 days after the last dose in the Open-Label Extension (OLE) study, are reported.
Arm/Group | Placebo; Bempedoic Acid | Bempedoic Acid; Bempedoic Acid | OLE Bempedoic Acid
All-Cause Mortality (participants affected / at risk) | 3/492 | 10/970 | 13/1462
Serious Adverse Events (participants affected / at risk) | 97/492 | 202/970 | 299/1462
Other Adverse Events (participants affected / at risk) | 108/492 | 201/970 | 309/1462
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo; Bempedoic Acid (N=492) | Bempedoic Acid; Bempedoic Acid (N=970) | OLE Bempedoic Acid (N=1462)
Coronary artery disease (Cardiac disorders) | 3 | 15 | 18
Angina pectoris (Cardiac disorders) | 5 | 9 | 14
Atrial fibrillation (Cardiac disorders) | 2 | 12 | 14
Angina unstable (Cardiac disorders) | 3 | 10 | 13
Acute myocardial infarction (Cardiac disorders) | 2 | 7 | 9
Myocardial ischaemia (Cardiac disorders) | 3 | 6 | 9
Myocardial infarction (Cardiac disorders) | 2 | 6 | 8
Cardiac failure (Cardiac disorders) | 0 | 5 | 5
Cardiac failure congestive (Cardiac disorders) | 3 | 2 | 5
Coronary artery stenosis (Cardiac disorders) | 0 | 4 | 4
Cardiac failure chronic (Cardiac disorders) | 0 | 3 | 3
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 6 | 9 | 15
Sepsis (Infections and infestations) | 2 | 4 | 6
Cellulitis (Infections and infestations) | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 2 | 2
Influenza (Infections and infestations) | 0 | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 2
Appendicitis (Infections and infestations) | 1 | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 1
Lymph node tuberculosis (Infections and infestations) | 0 | 1 | 1
Meningitis viral (Infections and infestations) | 0 | 1 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 6 | 8
Ischaemic stroke (Nervous system disorders) | 2 | 3 | 5
Cerebrovascular accident (Nervous system disorders) | 1 | 3 | 4
Syncope (Nervous system disorders) | 1 | 2 | 3
Carotid artery occlusion (Nervous system disorders) | 1 | 1 | 2
Cerebral infarction (Nervous system disorders) | 0 | 2 | 2
Presyncope (Nervous system disorders) | 1 | 1 | 2
Toxic encephalopathy (Nervous system disorders) | 1 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 1
External compression headache (Nervous system disorders) | 0 | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 6 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 4 | 1 | 5
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 5 | 8
Peripheral ischaemia (Vascular disorders) | 4 | 0 | 4
Aortic aneurysm (Vascular disorders) | 1 | 2 | 3
Hypertension (Vascular disorders) | 0 | 2 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 2
Angiodysplasia (Vascular disorders) | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 1
Temporal arteritis (Vascular disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 8 | 9
Chest pain (General disorders) | 1 | 4 | 5
Death (General disorders) | 0 | 2 | 2
Accidental death (General disorders) | 0 | 1 | 1
Brain death (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Hernia (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Vascular stent occlusion (General disorders) | 0 | 1 | 1
Vascular stent thrombosis (General disorders) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 1 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 6 | 8
Haematuria (Renal and urinary disorders) | 3 | 2 | 5
Ureterolithiasis (Renal and urinary disorders) | 0 | 2 | 2
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 1 | 6 | 7
Retinal artery occlusion (Eye disorders) | 0 | 1 | 1
Visual impairment (Eye disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 3 | 4
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2 | 3
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 1
Stress echocardiogram abnormal (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 1
Ultrasound ovary abnormal (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Adrenal cyst (Endocrine disorders) | 0 | 1 | 1
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1 | 1
Multiple endocrine neoplasia Type 1 (Congenital, familial and genetic disorders) | 0 | 1 | 1
Device malfunction (Product Issues) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 2
Acute left ventricular failure (Cardiac disorders) | 2 | 0 | 2
Anginal equivalent (Cardiac disorders) | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo; Bempedoic Acid (N=492) | Bempedoic Acid; Bempedoic Acid (N=970) | OLE Bempedoic Acid (N=1462)
Nasopharyngitis (Infections and infestations) | 33 | 86 | 119
Urinary tract infection (Infections and infestations) | 40 | 49 | 89
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 38 | 68
Upper respiratory tract infection (Infections and infestations) | 18 | 49 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03067441/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT03067441/SAP_001.pdf